CLINICAL TRIAL: NCT02880800
Title: Does the Use of Intravenous Patient Controlled Analgesia (IVPCA) Increase Opioid Consumption and Side Effects in Fast Track Orthopedic Procedures?
Brief Title: Does IVPCA Increase Opioid Consumption and Side Effects in Fast Track Orthopedic Procedures?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Naveed Siddiqui, Assistant professor, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 16-0098-A
Record Dates: First submitted 2016-08-17; First posted 2016-08-26 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Pain, Postoperative
Keywords: Analgesia, Patient-Controlled; Analgesics, Opioid; Drug-Related Side Effects and Adverse Reactions
MeSH Terms: conditions — Pain, Postoperative; Agnosia; Drug-Related Side Effects and Adverse Reactions | interventions — Morphine; Hydromorphone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Analgesia, patient controlled (Experimental): Patients will be given a patient controlled analgesia (PCA) pump containing a standard solution of either morphine or hydromorphone.
  Interventions: Drug: Morphine as IVPCA; Drug: Hydromorphone as IVPCA
- Analgesia, as per needed (Active Comparator): Patients will receive intravenous (IV) opioids as per needed.
  Interventions: Drug: Morphine; Drug: Hydromorphone

INTERVENTIONS:
Drug: Morphine as IVPCA — Morphine as IVPCA: Patients will be given a patient controlled analgesia (PCA) pump containing a standard solution of morphine as below:
  Morphine bolus 1mg with a lockout interval of 5 minutes, no background infusion and maximum 30 mg in 4 hours
  Other Names: Morphine
  Arms: Analgesia, patient controlled
Drug: Hydromorphone as IVPCA — Hydromorphone as IVPCA: Patients will be given a patient controlled analgesia (PCA) pump containing a standard solution of Hydromorphone as below:
  Hydromorphone bolus 0.2 mg with a lockout interval of 5 minutes and a maximum dose of 6 mg in 4 hours.
  Other Names: Dilaudid
  Arms: Analgesia, patient controlled
Drug: Morphine — IV opioids: Morphine 2 to 5 mg every 1h PRN (max. 20 mg/4h)
  Arms: Analgesia, as per needed
Drug: Hydromorphone — Hydromorphone 0.5 - 1 mg every 1h PRN (max. 4 mg/4h)
  Other Names: Dilaudid
  Arms: Analgesia, as per needed

SUMMARY:
The study aims to compare the use of intravenous patient controlled analgesia (IVPCA) versus the delivery of pain relief (per oral and intravenous (IV) medications as rescues analgesia) on an as needed basis within a well defined fast track protocol that includes multimodal analgesia for patients who are undergoing elective primary knee replacement surgery. The investigators assumed that with the multimodal analgesia regimen without the use of IVPCA will demonstrate decreased consumption of postoperative opioids, reduced incidence of opioids related side effects and decreased length of stay in the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 to 80 years old
* Provision of written informed consent
* Patients scheduled to undergo primary knee surgery included in the fast track protocol under regional anesthesia only
* Patients with Body Mass Index (BMI) between 18 to 34.9
* Patients with American Society of Anesthesiologists (ASA) physical status classification of 1 to 3

Exclusion Criteria:

* Patients on chronic (more than twice a week) opioid treatment including Tylenol #3, percocet, morphine, methadone, hydromorphone, fentanyl patch and other potent opioids
* Patients with language barrier or difficulty in communication in English
* Patients who are allergic to morphine and hydromorphone, fentanyl, gabapentin, celecoxib or acetaminophen
* Patients with increased risk for respiratory depression with intrathecal morphine (OSA, central apnea)
* Patients with documented Renal or hepatic impairment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Total amount of opioid consumption postoperatively | Every 24 hours for up to 48 hours after randomization

SECONDARY OUTCOMES:
Opioid related side effects. | Every 24 hours for up to 48 hours after randomization
  Opioid-related Symptom Distress Scale Questionnaire
Patient satisfaction | Once at 48 hours after randomization
  Patient satisfaction scale as below:
  1. Very dissatisfied
  2. Dissatisfied
  3. Slightly dissatisfied
  4. Slightly satisfied
  5. Satisfied
  6. Very satisfied
Pain scores measured at rest and movement | Every 12 hours for up to 48 hours after randomization
  Based on verbal analogue scale (VAS) scoring system (0-10), where score of 0 refers to no pain and a score of 10 refers to the worst pain imaginable
Length of stay in hospital | One week
  The total number of days the study patient was admitted in the hospital for a medical reason

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No